CLINICAL TRIAL: NCT00612924
Title: The Anaconda Endovascular Graft US FDA Phase II Clinical Study
Brief Title: The Vascutek AnacondaTM Stent Graft System Phase II IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo CVS (Industry)
Collaborators: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANA-006; G030036 (Other: FDA G030036)
Record Dates: First submitted 2008-01-22; First posted 2008-02-12 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Infrarenal Abdominal Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anaconda (Experimental)
  Interventions: Device: Anaconda Stent Graft System; Device: Anaconda ONE-LOK Stent Graft System

INTERVENTIONS:
Device: Anaconda Stent Graft System — Endovascular device
Device: Anaconda ONE-LOK Stent Graft System — Endovascular device

SUMMARY:
The Phase I safety study is now complete. FDA approval has been granted to proceed to Phase II. The primary objectives of the Phase II study is to assess the safety and effectiveness of the Anaconda Stent Graft System in subjects presenting with abdominal aortic aneurysm (AAA). The secondary objectives of this study are to assess additional clinical outcomes measurements associated with treatment of AAA using the Anaconda Stent Graft System

DETAILED DESCRIPTION:
Abdominal aortic aneurysms afflict a large number of patients in the United States and world-wide. The treatment of this disorder is based upon the concept of aneurysm repair prior to the presentation of symptoms or rupture. Thus aneurysm repair can be viewed as a prophylactic procedure embarked upon to prevent the disastrous complications of a ruptured aneurysm. The decision to treat an aneurysm electively is based upon a risk to benefit ratio. Treatment options include medical management of co-morbidities (hypertension, pulmonary disease, etc.) with observation of the aneurysm, open surgical aneurysm repair through a transabdominal or retroperitoneal approach, and endovascular aneurysm repair. The decision to intervene is based upon physician judgment. Once the decision to intervene is made, the mode of the intervention must be chosen. Although open surgical repair is more invasive and has been noted to have a higher morbidity and mortality(1;2) than most endovascular reports, few argue with the effectiveness of the procedure. To date, open surgical repair remains the gold standard of care for the aneurysm patient. Endovascular repair has several beneficial characteristics in comparison to an open surgical approach. They include the potential for decreased need for blood transfusions, shorter intensive care unit and total hospital stays, the lack of endotracheal intubation, to name a few. However, the procedure requires adequate imaging prior to graft placement and during the follow-up period, in addition to the availability of a trained team to ensure proper device placement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤ 85 years of age. Females must be non-pregnant, non-lactating, and not planning to become pregnant during the study period
* Females of childbearing potential must use acceptable methods of contraception, be at least one year post-menopausal or be surgically sterile
* Willing and able to comply with the 5 year follow-up period
* Willing to give informed written consent prior to enrollment
* Males with infrarenal AAA ≥ 4.5cm in diameter, or AAA growth ≥ 1.0cm/yr; females with infrarenal AAA ≥ 4.0cm in diameter, or AAA growth ≥ 1.0cm/yr
* Infrarenal AAA with a proximal neck diameter of 16.0 - 31.0mm (Anaconda Stent Graft System)
* Infrarenal AAA with a proximal neck diameter of 17.5 - 31.0mm (Anaconda ONE-LOK Stent Graft System)
* Infrarenal AAA with at least 15mm length of non-aneurysm proximal neck
* Infrarenal AAA with an angle of ≤ 60 degrees relative to the long axis of the aneurysm
* Iliac artery distal fixation sites ≥ 20mm in length
* Iliac artery distal fixation site ≤ 21mm in diameter
* Ability to preserve at least one hypogastric artery
* Femoral/iliac artery access vessels, size and morphology should be compatible with the appropriate introducer sheath (18 F, 20 F or 23 F).

Exclusion Criteria;

* Pregnant and lactating females or females of childbearing potential unless using acceptable method contraception
* Known sensitivity or allergy to nitinol or polyester
* Known allergy or intolerance of radiopaque contrast agents which cannot be pre-treated
* Thrombus, calcification, and/or plaque ≥ 2mm in thickness and/or ≥ 50% (180 degrees) continuous coverage of the vessel circumference in the intended fixation site
* Irregularly shaped calcification and/or plaque that may compromise the sealing and fixation at the proximal or distal fixation sites
* Ruptured or leaking AAA
* Mycotic or inflammatory AAA
* Genetic connective tissue disorder (i.e. Marfans or Ehlers-Danlos syndromes)
* Previous AAA repair
* Requires emergent AAA repair
* Concomitant thoracoabdominal aortic aneurysm
* Active systemic infection
* Myocardial infarction ≤10 weeks prior to procedure
* Aneurysm extends above renal arteries
* Dialysis dependent renal failure or creatinine > 2.5mg/dL
* Significant (>80%) renal artery stenosis not readily treatable
* End-stage chronic obstructive pulmonary disorder
* Patient is clinically and morbidly obese such that the required imaging would be prevented
* Patient has an uncorrectable bleeding abnormality
* Subject has other medical, social, or psychological problems that in the opinion of the investigator preclude them from receiving this treatment and the procedures and evaluations pre- and post- treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-04; Primary Completion 2013-07 (Actual); Study Completion 2017-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pregulman, MD, Study Director — Terumo Cardiovascular Systems Corporation
Locations (23):
- United States (18):
  - Arizona Heart Institute, Phoenix, Arizona
  - Central Arkansas Veteran's Hospital, Little Rock, Arkansas
  - Long Beach VA Healthcare System, Long Beach, California
  - University of Southern California Healthcare Consultation Ctr. II, Los Angeles, California
  - West Los Angeles VA Medical Centre, Los Angeles, California
  - Kaiser Permanente Hospital, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Florida Vascular Consultants, Maitland, Florida
  - Miller School of Medicine University of Miami, Miami, Florida
  - Southern Illinois Univ. School of Med., Springfield, Illinois
  - Indiana University Vascular Surgery, Methodist Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital Vascular and Endovascular Surgery, Boston, Massachusetts
  - Michigan Vascular Research Center, Flint, Michigan
  - University of Medicine and Dentistry of NJ, New Brunswick, New Jersey
  - Center for Vascular Awareness, Albany, New York
  - University of Buffalo surgeons, Inc., Buffalo, New York
  - Oregon Health and Science University, Portland, Oregon
  - Vascular and Transplant Specialist, Norfolk, Virginia
- Canada (5):
  - Peter Lougheed Center, Calgary, Alberta
  - St. Clare's Hospital, St. John's, Newfoundland and Labrador
  - London Health Science Center, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Johnston SC, Wilson CB, Halbach VV, Higashida RT, Dowd CF, McDermott MW, Applebury CB, Farley TL, Gress DR. Endovascular and surgical treatment of unruptured cerebral aneurysms: comparison of risks. Ann Neurol. 2000 Jul;48(1):11-9. doi: 10.1002/1531-8249(200007)48:13.3.co;2-m. PMID 10894211
- [Background] Greenberg RK, Lawrence-Brown M, Bhandari G, Hartley D, Stelter W, Umscheid T, Chuter T, Ivancev K, Green R, Hopkinson B, Semmens J, Ouriel K. An update of the Zenith endovascular graft for abdominal aortic aneurysms: initial implantation and mid-term follow-up data. J Vasc Surg. 2001 Feb;33(2 Suppl):S157-64. doi: 10.1067/mva.2001.111683. PMID 11174829
- See also: Company website — http://www.vascutek.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anaconda | ONE-LOK
Started | 101 | 94
Completed | 94 | 85
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Anaconda: The original protocol identified that the Anaconda™ Stent Graft System would be used throughout the current Phase II study. However, a modified device design became available during the course of the current Phase II study and is called the ONELOK™ Stent Graft System. As the modifications to the device design are considered minor, there are no expected differences in the anticipated safety or effectiveness of the device. The design changes relate primary to a uni-docking zone in the bifurcate body to maximize sizing compatibilities between the bifurcate body and the iliac limbs.
- Total: Total of all reporting groups
Arm/Group | Anaconda | ONE-LOK | Total
Number analyzed (Participants) | 101 | 94 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 86 | 79 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7.1) | 71 (7.3) | 71 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 85 | 82 | 167
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 34 | 74
  United States | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Successful Aneurysm Treatment
Description: defined as a composite endpoint of subjects who have successful delivery and deployment of the Anaconda™ Stent Graft at the initial procedure and at ≤365 days post-procedure and absence of:
  * Aneurysm growth ≥ 5 mm as evaluated by the core laboratory
  * Post-operative interventions to correct type I or III endoleaks
  * Conversion to open surgical repair
  * Failed patency of both limbs
  * Migration requiring secondary procedure or intervention
  * Significant fracture
  * Aneurysm rupture
Time Frame: 365 days
Population: In the ONE-LOK™ population, 85 subjects had efficacy endpoints and 9 subjects are missing due to withdrawal prior to 365-day follow-up. For the Anaconda population, 95 subjects had efficacy endpoints and 6 are missing data due to withdrawal prior to the 365-day follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Anaconda | ONE LOK
Number analyzed (Participants) | 95 | 85
percentage of patients | 90.9 [84.4 to 95.4] | 93.7 [88.5 to 97.9]

2. Secondary Outcome: Secondary Effectiveness, Technical Success
Description: Introduction and deployment of the Stent Graft in the absence of mortality, conversion to surgical repair, failed patency of both limbs, and evidence of a Type I or III endoleak through the first 24 hour post-operative period. The table below indicates the subjects who met the criteria for technical success based on Core Lab imaging evaluations.
Time Frame: 24 hours
Population: 151 subjects (81 Anaconda and 70 ONE-LOK) had imaging available for core lab review and determination of technical success.
Measure: Number; unit: participants
Arm/Group | Anaconda | ONE LOK | Total
Number analyzed (Participants) | 81 | 70 | 151
participants | 77 | 69 | 146

3. Primary Outcome: Freedom From Major Adverse Events
Description: The reported values represent the patients that did not experience a Major Adverse Event.
  Participants did NOT experience:
  * All-Cause Mortality
  * Myocardial Infarction (MI)
  * Cerebrovascular Accident (CVA)
  * Renal Failure
  * Respiratory Failure
  * Paralysis or Paraplegia, or
  * Bowel Ischemia
Time Frame: 30 days
Population: One Anaconda patient is not included in the analysis because their 30 day data was not reported.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Anaconda | ONE LOK
Number analyzed (Participants) | 100 | 94
percentage of patients | 96.6 [93.2 to 98.9] | 96.2 [92.3 to 98.6]

ADVERSE EVENTS:
Time Frame: 365 days
Arm/Group | Anaconda | ONE-LOK
Serious Adverse Events (participants affected / at risk) | 16/101 | 8/94
Other Adverse Events (participants affected / at risk) | 16/101 | 20/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anaconda (N=101) | ONE-LOK (N=94)
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Candiduria (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Death (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Device material issue (Injury, poisoning and procedural complications) | 1 | 0
Device Occlusion (Injury, poisoning and procedural complications) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Femoral Artery Aneurysm (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 2
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 3
Peripheral Artery Aneurysm (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 2
Peripheral embolism (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 1
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Renal artery occlusion (Renal and urinary disorders) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Injury, poisoning and procedural complications) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Serratia bacteraemia (Infections and infestations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Stent malfunction (Surgical and medical procedures) | 0 | 1
Stent removal (Surgical and medical procedures) | 1 | 0
Stent-graft endoleak (Injury, poisoning and procedural complications) | 3 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Thrombosis in device (Injury, poisoning and procedural complications) | 4 | 2
Transient ischemic attack (Nervous system disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 5 | 3
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anaconda (N=101) | ONE-LOK (N=94)
Hypertension (Vascular disorders) | 10 | 10
Stent-graft Endoleak (Injury, poisoning and procedural complications) | 6 | 10
Urinary Tract Infection (Infections and infestations) | 3 | 9
Procedural Pain (Injury, poisoning and procedural complications) | 8 | 7
Pyrexia (General disorders) | 5 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 8 | 4
Hypotension (Vascular disorders) | 7 | 3
Hypokalemia (Metabolism and nutrition disorders) | 6 | 3
Leukocytosis (Blood and lymphatic system disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less